CLINICAL TRIAL: NCT01080170
Title: The Effect of Aromatase Inhibitors on Cardiovascular Risk Factors in Women With Breast Cancer
Acronym: Silhouette
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Van Londen, Gijsberta, PI, University of Pittsburgh
Other Study IDs: PRO09060055; KL2RR024154-04 (NIH)
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: Aromatase Inhibitor; Anastrazole; Arimidex; Heart disease; Lipids; Body composition; Breast cancer.
MeSH Terms: conditions — Breast Neoplasms; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen serum samples. No further testing planned at the moment.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anastrazole: Newly diagnosed, non-metastatic, hormone-receptor positive breast cancer patients, who have undergone lumpectomy, have been advised to not require chemotherapy, but will need to undergo radiation therapy and will be initiating therapy with anastrazole.
- Control group - 2: Healthy controls.

SUMMARY:
This study explores how aromatase inhibitor therapy affects risk factors for heart disease in postmenopausal women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory women (aged 60-75), with a new diagnosis of nonmetastatic, hormone-receptor positive breast cancer, having undergone lumpectomy. They will not need chemotherapy and will have been prescribed but not yet started anastrazole. All will need a course of radiation therapy as part of usual care. Participants are instructed not to change their physical activity or eating habits over the period of the study.

Comparisons are:

* Identical to the cases except they are hormone-receptor negative and don't need hormonal therapy.
* Healthy controls.

Exclusion Criteria:

* Nicotine usage
* Metastatic breast cancer
* Need for chemotherapy
* AI other than anastrazole
* Usage of steroids (equivalent of equal then or more than 7.5 mg prednisone x 3 months)
* Clinically significant abnormality of thyroid function
* Treatment with gonadal hormone replacement therapy within last 3 years
* Status post unilateral/bilateral surgical oophorectomy
* Having experienced a medical event, which may confound study outcomes [e.g. heart attack, stroke, cancer (metastatic or newly diagnosed within last 5 years, except for non-melanoma skin cancer and breast), lupus, rheumatoid arthritis, chronic inflammatory disease]
* Medication-dependent diabetes mellitus or hypercholesterolemia.
* Gastric surgery
* Weight loss medication (prescription or over the counter)

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients will be recruited via the Magee Breast Cancer Program of the Cancer Center at the University of Pittsburgh Medical Center. Healthy controls will be recruited via registries.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Body Composition | 12 months

SECONDARY OUTCOMES:
Lipids | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Department of Medicine., Pittsburgh, Pennsylvania, United States